CLINICAL TRIAL: NCT01506947
Title: A Prospective, Non-randomised, Single-arm, Open-Label Pilot Clinical Study Evaluating the Effect of PTH Lowering on Erythropoietin Consumption in Calcitriol-Resistant Patients
Brief Title: A Pilot Clinical Study Evaluating the Effect of Parathyroid Hormone (PTH) Lowering On Erythropoietin Consumption in Calcitriol-Resistant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W12-645
Record Dates: First submitted 2011-12-28; First posted 2012-01-10 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Moderate to Severe Secondary Hyperparathyroidism; Stage 5 Chronic Kidney Diseases
Keywords: Hemodialysis; Chronic kidney disease; Secondary hyperparathyroidism,
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary | interventions — paricalcitol; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paricalcitol (Experimental): Participants received paricalcitol intravenously during hemodialysis until serum intact parathyroid hormone (iPTH) levels were below 150 pg/mL or for up to 6 months. Paricalcitol dose was based on iPTH levels and was titrated to maintain iPTH levels between 150-300 pg/mL.
  Participants may have also received routine darbepoetin alfa to treat anemia.
  Interventions: Drug: Paricalcitol; Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Paricalcitol — Paricalcitol was administered by intravenous bolus. The initial dose was calculated according to the following formula:
  [Paricalcitol (µg) = iPTH (pg/mL) / 80]. Subsequent doses were determined based on iPTH, calcium and phosphorus levels.
  Other Names: ABT-358; Zemplar
Drug: Darbepoetin alfa — Routine darbepoetin alfa use was allowed when transferrin saturation (TSAT) was ≥ 20% and ferritin ≥ 200 μg/L, and hemoglobin level < 11.5 g/dL. The initial dose was 0.25 to 0.75 µg/kg/week, and the maintenance dose was 0.13 to 0.35 µg/kg/week. Target hemoglobin level was between 10 to 11.5 g/dL.

SUMMARY:
To evaluate the effect of PTH lowering on erythropoietin consumption in calcitriol-resistant patients with stage 5 chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria: A subject will only be included if all the following entry criteria are met:

* Patients ≥ 18 years of age
* Stage 5 chronic kidney disease (CKD) patients receiving hemodialysis and with moderate to severe secondary hyperparathyroidism (SHPT)
* Patients with anemia due to renal insufficiency but who are iron replete:; Transferrin saturation (TSAT) > 20% and Ferritin levels > 200 ng/mL and requiring treatment with erythropoietin (EPO)
* Patients with vitamin B levels > lower limit of normal (LLN) and folic acid levels > LLN
* Patients treated only with intravenous calcitriol for at least 6 months
* Patients with serum intact parathyroid hormone (iPTH) level > 500 pg/mL
* Patients with calcium phosphate product (Ca × PO4) < 65 mg²/dL²
* Patients willing to sign "written informed consents" before participating in any the study related activity.
* Patients with phosphorus levels < 6.5 mg/dL and calcium levels < 11.2 mg/dL

Exclusion Criteria:

A subject will be excluded from the study if he/she meets any of the following criteria:

* Patients who have known hypersensitivity and/or toxicity to vitamin D metabolites and/or to paricalcitol and/or to other product ingredients.
* Patients who have participated in a clinical study within the last month.
* Patients whose previous concomitant medication and laboratory data for 6 months prior to the baseline visit are not available.
* Patients with known contraindication to selective Vitamin D receptor activators (VDRAs) according to the Summary of Product Characteristics (SmPC).
* Pregnancy, breast-feeding or planning a pregnancy within next 6 months after enrollment. Sexually active female patients not accepting appropriate contraceptive methods during the course of the study will also be excluded.
* Hypertensive and diabetic patients who are not on an optimal and steady medication regimen for more than 30 days.
* Patients with microcytic (mean corpuscular volume [MCV] < 80 fL) and macrocytic (MCV > 100 fL) anemia at screening that may be caused by diseases such as for microcytic anemias - Iron Deficiency, Thalassemias, Anemia of Chronic Disease, Copper Deficiency, Zinc poisoning, Sideroblastic Anemia, macrocytic anemias -ethanol abuse, myelodysplastic syndromes, acute myeloid leukemias, reticulocytosis, drug induced anemia, liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-05-10 (Actual); Primary Completion 2016-04-07 (Actual); Study Completion 2016-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Gücük, MD, Study Director — AbbVie

REFERENCES:
- [Background] Poordad F, Landis CS, Asatryan A, Jackson DF 3rd, Ng TI, Fu B, Lin CW, Yao B, Kort J. High antiviral activity of NS5A inhibitor ABT-530 with paritaprevir/ritonavir and ribavirin against hepatitis C virus genotype 3 infection. Liver Int. 2016 Aug;36(8):1125-32. doi: 10.1111/liv.13067. Epub 2016 Feb 3. PMID 26778412
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 7 centers in Turkey.
Period: Overall Study
Arm/Group | Paricalcitol
Started | 65
Completed | 49
Not Completed | 16
Not completed — Lost to Follow-up | 7
Not completed — Adverse Event | 5
Not completed — Death | 1
Not completed — Did Not Meet Eligibility Criteria | 3

BASELINE CHARACTERISTICS:
Population: The per-protocol analysis set which included participants who completed the study according to the protocol. One patient was enrolled into the study under protocol version 1.0 and was not included in the per-protocol analysis set due to subsequent major changes to the protocol.
Arm/Group | Paricalcitol
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Erythropoietin Dose Per Visit
Description: The requirement of erythropoietin (EPO) treatment to maintain serum hemoglobin levels between 10 to 11.5 g/dL during the study was assessed by analysis of the dose of darbepoetin alfa used at baseline and during each month of the study. The mean EPO dosage per injection for each study month is reported.
Time Frame: Baseline and Months 1, 2, 3, 4, 5 and 6
Population: Per-protocol analysis set with EPO dosage available at all visits.
Measure: Mean (Standard Deviation); unit: µg
Arm/Group | Paricalcitol
Number analyzed (Participants) | 45
µg
  Baseline | 35.8 (15.0)
  Month 1 | 22.2 (20.0)
  Month 2 | 22.7 (21.3)
  Month 3 | 4.7 (4.5)
  Month 4 | 7.2 (6.2)
  Month 5 | 17.3 (19.5)
  Month 6 | 21.8 (19.7)

2. Secondary Outcome: Mean Scores of Short Form Health Survey 36 (SF-36) Questionnaire
Description: The Medical Outcome Study Short Form 36-Item Health Survey (SF-36) is a self-administered questionnaire that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains. The domains include physical (physical functioning, role limitations due to physical health (role-physical), general health perceptions and pain) and mental domains (energy/fatigue (vitality), social functioning, emotional well-being (mental health), and role limitations due to emotional problems (role emotional)). The individual domain scores are calculated and transformed to range from 0 to 100, with higher scores indicating a better level of functioning.
Time Frame: Baseline and Month 6
Population: Per-protocol analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paricalcitol
Number analyzed (Participants) | 48
units on a scale
  Physical Function - Baseline | 51.7 (26.3)
  Physical Function - Month 6 | 51.5 (30.1)
  Role Physical - Baseline | 38.5 (45.2)
  Role Physical - Month 6 | 44.3 (46.5)
  Role Emotional - Baseline | 52.8 (46.0)
  Role Emotional - Month 6 | 54.2 (47.0)
  Vitality - Baseline | 47.4 (16.5)
  Vitality - Month 6 | 45.2 (17.0)
  Mental Health - Baseline | 54.5 (12.6)
  Mental Health - Month 6 | 52.7 (15.2)
  Social Functioning - Baseline | 59.6 (20.7)
  Social Functioning - Month 6 | 55.5 (26.3)
  Pain - Baseline | 61.3 (26.6)
  Pain - Month 6 | 60.5 (25.0)
  General Health - Baseline | 47.0 (16.9)
  General Health - Month 6 | 44.4 (22.3)

3. Secondary Outcome: Mean Intact Parathyroid Hormone (iPTH) Level at Baseline and Month 6
Time Frame: Baseline and Month 6
Population: Per-protocol analysis set with available data at each time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Paricalcitol
Number analyzed (Participants) | 48
pg/mL
  Baseline | 918.0 (585.9)
  Month 6: number analyzed (Participants) | 46
  Month 6 | 692.5 (413.4)

4. Secondary Outcome: Mean Calcium Level at Baseline and Month 6
Time Frame: Baseline and Month 6
Population: Per-protocol analysis set with available data at each time point.
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Paricalcitol
Number analyzed (Participants) | 48
mg/mL
  Baseline | 8.81 (0.95)
  Month 6: number analyzed (Participants) | 46
  Month 6 | 9.29 (0.86)

5. Secondary Outcome: Mean Phosphorus Level at Baseline and Month 6
Time Frame: Baseline and Month 6
Population: Participants who completed the study with available data at each time point.
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Paricalcitol
Number analyzed (Participants) | 48
mg/mL
  Baseline | 4.87 (1.11)
  Month 6: number analyzed (Participants) | 46
  Month 6 | 5.47 (1.22)

6. Secondary Outcome: Mean Alkaline Phosphatase Level at Baseline and Month 6
Time Frame: Baseline and Month 6
Population: Per-protocol analysis set with available data at each time point.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Paricalcitol
Number analyzed (Participants) | 48
U/L
  Baseline | 225.7 (170.1)
  Month 6: number analyzed (Participants) | 46
  Month 6 | 172.9 (147.6)

7. Secondary Outcome: Vitamin B12 Levels
Description: Vitamin B12 levels were categorized according to the following laboratory reference ranges:
  Low: < 200 pg/mL Normal: 200 - 950 pg/mL High: > 950 pg/mL
Time Frame: Baseline and month 6
Population: Per-protocol analysis set with available data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline | Month 6
Number analyzed (Participants) | 48 | 46
Participants
  Low | 2 | 0
  Normal | 13 | 22
  High | 33 | 24

8. Secondary Outcome: Folic Acid Levels
Description: Folic acid levels were categorized according to the following laboratory reference ranges:
  Low: < 4.6 ng/mL Normal: 4.6 - 18.7 ng/mL High: > 18.7 ng/mL
Time Frame: Baseline and month 6
Population: Per-protocol analysis set with available data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline | Month 6
Number analyzed (Participants) | 48 | 46
Participants
  Low | 1 | 4
  Normal | 25 | 25
  High | 22 | 17

9. Secondary Outcome: Mean High Sensitivity C-reactive Protein (hsCRP) Level at Baseline and Month 6
Time Frame: Baseline and Month 6
Population: Per-protocol analysis set with available data at each time point.
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Paricalcitol
Number analyzed (Participants) | 48
mg/mL
  Baseline | 11.8 (14.1)
  Month 6: number analyzed (Participants) | 46
  Month 6 | 14.4 (20.7)

10. Secondary Outcome: Mean Fibroblast Growth Factor-23 (FGF-23) Level at Baseline and Month 6
Time Frame: Baseline and Month 6
Population: Per-protocol analysis set with available data at each time point.
Measure: Mean (Standard Deviation); unit: kRU/L
Arm/Group | Paricalcitol
Number analyzed (Participants) | 46
kRU/L
  Baseline | 6267 (5967)
  Month 6: number analyzed (Participants) | 44
  Month 6 | 11340 (13450)

11. Secondary Outcome: Number of Participants With Adverse Events
Description: Serious adverse events were any adverse events meeting any of the following criteria:
  * An event that resulted in the death of a participant;
  * An event that, in the opinion of the investigator, would have resulted in immediate fatality if medical intervention had not been taken (life-threatening);
  * Resulted in an admission to the hospital for any length of time or prolonged hospital stay;
  * An anomaly detected at or after birth, or any anomaly that results in fetal loss;
  * An event that resulted in a condition that substantially interfered with the activities of daily living;
  * An important medical event that may not be immediately life-threatening or result in death or hospitalization, but based on medical judgment may have jeopardized the participant and may have required medical or surgical intervention to prevent any of the outcomes listed above.
  Adverse events were assessed by the investigator for possible relationship to study drug.
Time Frame: From the time of study drug administration until 4 weeks after the discontinuation of the study drug; up to 7 months.
Population: The safety population included all participants who enrolled.
Measure: Number; unit: participants
Arm/Group | Paricalcitol
Number analyzed (Participants) | 65
participants
  Non-serious adverse events | 9
  Serious adverse events | 11
  Treatment-related adverse events | 0
  Fatal adverse events | 3

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Paricalcitol
Serious Adverse Events (participants affected / at risk) | 11/65
Other Adverse Events (participants affected / at risk) | 1/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol (N=65)
Nephrectomy (Surgical and medical procedures) | 1
Asthenia (General disorders) | 2
Fatigue (General disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Parathyroidectomy (Surgical and medical procedures) | 1
Renal transplant (Surgical and medical procedures) | 2
Soft tissue infection (Infections and infestations) | 1
Pyrexia (General disorders) | 2
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Lung infection (Infections and infestations) | 1
Chest Pain (General disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Palpitations (Cardiac disorders) | 2
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Acute Respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac valve disease (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Respiratory Tract Infection (Infections and infestations) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Somnolence (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Stools watery (Gastrointestinal disorders) | 1
Faeces discoloured (Gastrointestinal disorders) | 1
Haemoglobin decreased (Investigations) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2
Haemoconcentration (Blood and lymphatic system disorders) | 1
Haemoglobin increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol (N=65)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1
Nasopharyngitis (Infections and infestations) | 1
Arteriovenous fistula (Vascular disorders) | 1
Headache (Nervous system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Dizziness (Nervous system disorders) | 1
Chest pain (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pain (General disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.